CLINICAL TRIAL: NCT04811183
Title: Pharmaceutical Consultation and Exchange Between the Pharmacy and the Hospital
Acronym: EPHET
Status: Withdrawn | Type: Observational
Why Stopped: No participants enrolled
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL21_0197
Record Dates: First submitted 2021-03-19; First posted 2021-03-23 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Diabetes
Keywords: pharmaceutical consultations; adherence
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Experimental group: Adult patients hospitalized with diabetes and polymedicated. Selected to benefit from a pharmaceutical consultation before their return home.
  Interventions: Behavioral: Pharmaceutical consultation

INTERVENTIONS:
Behavioral: Pharmaceutical consultation — Selection of patients for a pharmaceutical consultation with collection of non-opposition and scheduling of telephone interviews or by teleconsultations at one week after hospitalization.
  Data collection through interviews using a telephone questionnaire (or by teleconsultation) one week after consultation. Elements on knowledge and adherence of treatment will be collected.

SUMMARY:
Investigators hypothesize that the implementation of a hospital pharmacy consultation and the transmission of its report to pharmacies may improve knowledge, adherence and encourage the development of pharmacist medication reviews. A before-and-after study of the implementation of pharmaceutical consultations will allow the investigators to evaluate the validity of the hypothesis.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient admitted in the endocrinology service for a type 2 Diabetes who has more than 5 concomitant treatments
* Adult patient that is being discharged for a return home
* Good comprehension of French

Exclusion Criteria:

* Bad comprehension of French

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patient admitted in the endocrinology service for a type 2 Diabetes who has more than 5 concomitting treatments, on the way to returning home.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2023-06-23 (Actual); Primary Completion 2023-06-23 (Actual); Study Completion 2023-06-23 (Actual)

PRIMARY OUTCOMES:
Evolution in the knowledge about the patient's condition | One week
  Treatment knowledge, knowledge about the pathology and knowledge of hygienic and dietary measures will be assessed with a questionnaire giving a score from 0 to 2 -the higher the score, the better the outcome-.
  Comparison of the knowledge of the treatment between the first questionnaire conducted during the pharmaceutical consultation and the second questionnaire one week after the consultation.
  Statistical evaluation by comparative tests between the two questionnaires.
Evolution in the adherence | One week
  Evaluation of the patient's adherence to his treatment through a questionnaire giving a score between 0 to 6 -the higher the score, the better the outcome-. Comparison of the scores between the first questionnaire conducted during the pharmaceutical consultation and the second questionnaire one week after the consultation.
  Statistical evaluation by comparative tests between the two questionnaires.

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Louis Pradel, Bron, France